CLINICAL TRIAL: NCT00522834
Title: A Randomized, Double-blind, Phase 3 Trial of Elesclomol (STA-4783) in Combination With Paclitaxel Versus Paclitaxel Alone for Treatment of Chemotherapy-Naïve Subjects With Stage IV Metastatic Melanoma (SYMMETRY)
Brief Title: Elesclomol (STA-4783) With Paclitaxel Versus Paclitaxel Alone in Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4783-08
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Melanoma
Keywords: melanoma; oncology; Stage IV Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — elesclomol; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Elesclomol (STA-4783) in Combination With Paclitaxel
  Interventions: Drug: Elesclomol (STA-4783)
- 2 (Other): Paclitaxel alone
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Elesclomol (STA-4783) — 213 mg/m2 Elesclomol (STA-4783) plus 80 mg/m2 paclitaxel administered intravenously once a week for the first 3 weeks of a 4 week cycle. Number of cycles: Until progression or unacceptable toxicity develops
  Arms: 1
Drug: Paclitaxel — 80 mg/m2 paclitaxel alone administered intravenously once a week for the first 3 weeks of a 4 weeks cycle. Number of cycles: Until progression or unacceptable toxicity develops
  Arms: 2

SUMMARY:
"Elesclomol (STA-4783), N-malonyl-bis (N'-methyl-N'-thiobenzoylhydrazide) is a new chemical entity with a novel structure. STA-4783 induces an oxidative stress response in cells. This response is characterized by increased production of gene families that protect against different cellular stresses, including excessive heat, the presence of reactive oxygen species such as oxygen radicals, or the presence of heavy metals.

Subjects will participate in up to 2 weeks of screening during which time they will complete all screening procedures. Eligible subjects who have not received any prior cytotoxic chemotherapeutic agent for melanoma will be randomized in a 1:1 ratio to receive either STA-4783 213 mg/m2 in combination with paclitaxel 80 mg/m2 or paclitaxel 80 mg/m2 alone.

One treatment cycle will consist of weekly treatments for 3 weeks, followed by a 1-week rest period. Cycles will be repeated every 4 weeks until disease progression. Tumor assessments will be performed every 8 weeks from the date of randomization or sooner if the Investigator suspects progression has occurred based on clinical signs and symptoms. "

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic (Stage IV) melanoma of cutaneous origin
* ECOG performance status of <=2
* Measurable disease according to modified RECIST
* Life expectancy of greater than 12 weeks
* LDH <= 2.0 x ULN
* Clinical lab values within protocol parameters.
* At least 18 years old and able and willing to provide informed consent to participate

Exclusion Criteria:

* Previous cytotoxic chemotherapy treatment for melanoma
* Received more than one regimen of immunotherapy, kinase inhibitor, biologic therapy, vaccine or investigational non-chemotherapeutic treatment for melanoma.
* Presence of brain metastases
* Presence or history (<= 5 years) of a second malignancy other than nonmelanoma skin cancer or cervical carcinoma in situ
* Female subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | June 2009

SECONDARY OUTCOMES:
Overall Survival | December 2009
Objective response rate | December 2009
Clinical benefit rate | December 2009
Duration of objective response | December 2009
Safety | December 2009
Pharmacokinetics | December 2009

CONTACTS AND LOCATIONS:
Locations (101):
- United States (61):
  - Arizona Cancer Center, Tucson, Arizona
  - Winthrop P. Rockefeller Cancer Institute, Little Rock, Arkansas
  - University of California San Diego Moores UCSD Cancer Center, La Jolla, California
  - University of California, San Diego, La Jolla, California
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - Jonsson Comprehensive Cancer Center Univ. of California Los Angeles, Los Angeles, California
  - Pacific Medical Center Research Institute, San Francisco, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Anschutz Cancer Pavillion University of Colorado, Aurora, Colorado
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Univ. of Miami Hospital and Clinics, Miami, Florida
  - MD Anderson Cancer Center, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Rush University Hospital, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Joliet Oncology/Hematology Associates, LTD, Joliet, Illinois
  - Oncology Specialists, S.C., Niles, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Wayne State University, Detroit, Michigan
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Ellis Fischels Cancer Center, Columbia, Missouri
  - Southeast Nebraska Hematology/Oncology, Lincoln, Nebraska
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Health Research - Mountainside Hospital, Montclair, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Monter Cancer Center North Shore Hospital, Lake Success, New York
  - Weill Medical College of Cornell University - Division of Hematology and Medical Oncology, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - Stony Brook University Medical Center- Cancer Center, Stony Brook, New York
  - UNC School of Medicine - Division of Hematology/Oncology, Chapel Hill, North Carolina
  - Carolina Hematology & Oncology Associates, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - Brody School of Medicine at East Carolina State University, Greenville, North Carolina
  - Derrick L. Davis Regional Cancer Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University., Columbus, Ohio
  - Mark H. Zangmeister Cancer Center, Columbus, Ohio
  - Providence Cancer Center Clinical Trials, Portland, Oregon
  - St. Luke's Cancer Center, Bethlehem, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Cancer Pavilion, Pittsburgh, Pennsylvania
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Texas Oncology, PA, Dallas, Texas
  - San Antonio Cancer Institute, San Antonio, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Australia (11):
  - Lismore Base Hospital, Cancer Care & Haematology Unit, Lismore, New South Wales
  - Newcastle Melanoma Unit - Calvary Mater Newcastle, Waratah, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Redcliffe Hospital, Redcliffe, Queensland
  - Princess Alexandra Hospital, Wooloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Adelaide Cancer Centre Medical Oncology, Adelaide
  - Patricia Ritchie Centre for Cancer Care and Research, Mater Hospital, North Sydney
  - The Tweed Hospital, Tweed Heads
  - Department of Medical Oncology, Westmead Hospital, Westmead
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - QE II Health Sciences Center, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Cross Cancer Institute, Edmonton
  - Princess Margaret Hospital, Toronto
- Germany (10):
  - Vivantes Klinikum Im Friedrichshain, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Elbe-Klinikum Buxtehude, Buxtehude
  - Universität zu Köln, Cologne
  - University Frankfurt, Frankfurt am Main
  - University of Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Würzburg, Würzburg
- VA Medical Center, San Juan, Puerto Rico
- Romania (6):
  - County Hospital Brasov - Oncology Department, Brasov
  - Oncology Institute "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Clinical County Hospital " Alexandru Simionescu" Hunedoara, Hunedoara
  - Center of Medical Oncology, Iași
  - Clinical County Hospital Sibiu, Sibiu
  - Oncology- Chemotherapy Clinic - Emergency Municipal Clinical Hospital, Timișoara
- Spain (4):
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de la Princessa Servicio de Oncología Médica, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Virgen de la Salud - Servicio de Oncología Médica Ciclos, Toledo
- United Kingdom (3):
  - Oncology Centre Addenbrookes's Hospital, Cambridge
  - Northern Centre for Cancer Treatment Newcastle General Hospital, Newcastle upon Tyne
  - Dorset Cancer Centre Poole Hospital NHS Foundation Trust, Poole

REFERENCES:
- [Derived] O'Day SJ, Eggermont AM, Chiarion-Sileni V, Kefford R, Grob JJ, Mortier L, Robert C, Schachter J, Testori A, Mackiewicz J, Friedlander P, Garbe C, Ugurel S, Collichio F, Guo W, Lufkin J, Bahcall S, Vukovic V, Hauschild A. Final results of phase III SYMMETRY study: randomized, double-blind trial of elesclomol plus paclitaxel versus paclitaxel alone as treatment for chemotherapy-naive patients with advanced melanoma. J Clin Oncol. 2013 Mar 20;31(9):1211-8. doi: 10.1200/JCO.2012.44.5585. Epub 2013 Feb 11. PMID 23401447